CLINICAL TRIAL: NCT05401890
Title: Association Between Serum Ferritin Level and Severity of Liver Disease and Development of HCC in Cirrhotic Patients.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hala Hany Faheem Fadl allh, Doctor, Assiut University
Other Study IDs: Serum ferritin level
Record Dates: First submitted 2022-05-30; First posted 2022-06-02 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-05

CONDITIONS: HCC

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Association between serum ferritin level and severity of liver disease and development of HCC in cirrhotic patients .

DETAILED DESCRIPTION:
th leading cause of cancer mortality worldwide, with an estimated 841,000 (9.3 cases per 100,000 person-years) and 782,000 deaths (8.5 deaths per 100,000 person-years) in 2018.(Bray F et al., 2018) In Egypt, it represents the fourth common cancer and the leading cause of mortality- and morbidity-related cancer .(Akinyemiju T, et al.T 2017) Many hospital based studies reported increasing the incidence of HCC The reason for increased incidence could be attributed to improvement in screening programs and diagnostic tools, increasing the survival rate of cirrhotic patients that increases the chance of developing HCC . (Ibrahim AS, et al 2014) Because the early stage disease is usually asymptomatic, approximate half of patients are diagnosed at an advanced stage. Many biomarkers, such as α-fetoprotein (AFP) have already been used to screen for HCC and choose the best treatment on an individual status. However, these biomarkers are not sufficient to predict prognosis accurately. (Kabbach G, 2015) Ferritin, as a soluble iron-storage protein, participates in iron metabolism and accumulation, which directly damage DNA and proteins by generating reactive species and cause apoptosis through activation of the caspase cascade and hyperoxidation of fatty chains(Miyanishi K et al., 2019). Additionally, it is believed to be responsible for enhanced production of collagen and liver fibrosis . (Wang W et al., 2010) Elevated serum ferritin is frequently observed among patients with liver injury, regardless of etiology. (Wong K, Adams PC, 2006) However, whether ferritin is associated with incident liver cancer remains unclear. On one hand, previous clinical and epidemiologic studies show that serum ferritin may be correlated with liver cancer risk. For example, a recent meta-analysis including nine studies showed that higher serum ferritin was associated with 1.5-fold increases in risk of liver cancer. (Tran KT et al., 2019) On the other hand, the serum ferritin levels were associated with liver cancer among HCV+ men but not women in a Japanese cohort study. (Uchino K et al 2016 ) Moreover, no study has evaluated association between serum ferritin levels and the severity of hepatic decompensation in cirrhotic patients. Therefore, we will carry out a case-control study in Al Rajhy Liver Hospital, Assiut University, to examine the association between serum ferritin concentration and the incidence of HCC and severity of hepatic impairment in subjects with liver cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with liver cirrhosis of both sexes with and without HCC regardless of the aetiology of chronic liver disease

Exclusion Criteria:

* Patients less than 18 years Previously treated HCC patients with no evidence of recurrence or residual activity Subjects who had received blood transfusions or iron supplements during the previous 3 months.

Other conditions associated with elevated serum ferritin e.g., malignancy other than HCC, iron overload syndromes, autoimmune disorders, chronic excess alcohol consumption and acute and chronic infections.

Patients who will refuse to give a written consent, will be excluded from our study

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with liver cirrhosis of both sexes with and without HCC regardless of the aetiology of chronic liver disease
Sampling Method: Non-Probability Sample
Enrollment: 102 (Estimated)
Dates: Start 2022-08-01 (Estimated); Primary Completion 2023-08-01 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
Association between serum ferritin level and severity of liver disease and development of HCC in cirrhotic patients . | One year
  The relation between serum ferritin level and severity of liver disease and development of HCC in cirrhotic patients

REFERENCES:
- [Result] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. (2018) 68:394-424.doi: 10.3322/caac.21492 . Akinyemiju T, Abera S, Ahmed M, Alam N, Alemayohu MA, Allen C, et al.The burden of primary liver cancer and underlying etiologies from 1990 to 2015 at the global, regional, and national level. JAMA Oncol. 2017;3:1683-91.https://doi.org/10.1001/jamaoncol.2017.3055. Ibrahim AS, Khaled HM, Mikhail NN, Baraka H, Kamel H. Cancer incidence in Egypt: results of the national population-based cancer registry program. J Cancer Epidemiol. 2014;2014:437971.https://doi.org/10.1155/2014/437971 . Kabbach G, Assi HA, Bolotin G, et al. Hepatobiliary Tumors: Update on Diagnosis and Management. J Clin Transl Hepatol 2015;3:169-81. Miyanishi K, Tanaka S, Sakamoto H, Kato J. The role of iron in hepatic inflammation and hepatocellular carcinoma.Free Radic. Biol. Med.2019;133: 200-5. Wang W, Knovich MA, Coffman LG, Torti FM, Torti SV. Serum ferritin: past, present and future.Biochim. Biophys. Acta2010;1800:760-9. Wong K, Adams PC. The diversity of liver diseases among outpatient referrals for an elevated serum ferritin.Can. J. Gastroenterol.2006;20:467-70. Tran KT, Coleman HG, McCain RS, Cardwell CR. Serum biomarkers of iron status and risk of primary liver cancer: a systematic review and meta-analysis.Nutr. Cancer2019;71: 1365-73. Uchino K, Tateishi R, Fujiwara Net al. Impact of serum ferritin level on hepatocarcinogenesis in chronic hepatitis C patients.Hepatol. Res.2016;46: 259-68.